CLINICAL TRIAL: NCT05459441
Title: Efficacy and Safety Evaluation of Percutaneous Ommaya Capsule Injection of Autologous Bi-dimensional Specific T Cells in the Treatment of Glioma and in Combination With Pemetrexed in the Treatment of Brain/Meningeal Metastases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-IIT-004-F01
Record Dates: First submitted 2022-06-24; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-02

CONDITIONS: Glioma; Brain Metastases
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: Single center prospective clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of glioma (Experimental): For patients with glioma, after the patient's general condition was stable, contraindications were excluded and RAK cells were injected into Ommaya sac.
  Interventions: Biological: Autologous progenitor expansion -T
- Treatment of brain metastases (Experimental): For patients with brain/meninges metastasis, Ommaya capsule was placed subcutaneously after puncture under local anesthesia. Two days after surgery, chemotherapy was started when the intracranial pressure was stable and the condition was stable, and the conjunctivitis was eliminated. Intracapsular injection of autoimmune cells was started in the second week after chemotherapy.
  Interventions: Biological: Autologous progenitor expansion -T; Drug: pemetrexed

INTERVENTIONS:
Biological: Autologous progenitor expansion -T — After the completion of RAK cell culture, RAK cells were slowly injected into the tumor cavity through Ommaya capsule for no less than 10 minutes, each time about 1.0-4.0 108/4 mL, once a week,3 times as a course of treatment. Il-2 (500,000 units/capsule) was injected into the tumor cavity through Ommaya reservoir every other day after the injection of RAK cells In other words, the day of RAK cell injection was the first day, and the third and fifth days were respectively injected. Then, about LML of sac fluid was pumped back before each injection to observe the growth of RAK cells in the tumor cavity. Il-2 was dissolved with LML normal saline, and the fluid storage sac was pressed 3-5 times after injection to make the sac fluid and IL-2 fully mixed.
Drug: pemetrexed — For patients with brain metastasis from solid tumor that met the inclusion conditions, the Ommaya capsule was placed 2 days later, and the maximum tolerated dose of pemetrexed intrathecal chemotherapy was injected intravaginally at 10mg according to the general situation of the patients and the results of the previous study.
  Arms: Treatment of brain metastases

SUMMARY:
Cerebral metastases are common intracranial tumor, its incidence increased year by year, in recent years, although the whole brain radiation therapy, surgical resection, stereotactic radiosurgery treatment, targeted drugs, and other comprehensive treatment in patients with symptoms of mitigation and the extension of survival has played a positive role, but due to individual differences, treatment in patients with poor compliance were a lot of factors, Further treatment of brain metastases after conventional treatment requires the assistance and cooperation of clinical multi-disciplines. To evaluate the efficacy and safety of percutaneous Ommaya capsule injection of autologous bi-dimensional specific T cells in the treatment of glioma and combined with pemetrexed in the treatment of brain/meningeal metastasis. Using translational research techniques and means, to find molecular indicators related to clinical prognosis and outcome, establish the clinical use standard of this holistic treatment technology, and popularize it in multi-centers.

ELIGIBILITY:
Inclusion Criteria:

1. Clear diagnosis of glioma; The pathological diagnosis of the primary lesion is clear, and the intracranial lesion can be diagnosed as intracranial metastasis by clinical, cerebrospinal fluid and imaging diagnosis according to the standards of the European Society of Neuro-Oncology - European Society of Medical Oncology (EANo-ESMO).
2. Patients with glioma and solid tumor with brain metastasis who have relapsed after surgery, whole brain radiotherapy or chemotherapy, or who are intolerant and not suitable for surgery or radiotherapy, and who are determined by clinicians to no longer benefit from systemic chemotherapy;
3. Surgical indications for Ommaya capsule implantation;
4. Age ≥18 years old and ≤80 years old, regardless of gender;
5. ECOG score for general physical condition is 0 ~ 2;
6. The expected survival time is at least 1 month;
7. WBC≥3.0×109/L, Hb≥90g/L, PLT≥75×109/L at baseline upon enrollment;
8. Liver and kidney function are basically normal A) Liver: total bilirubin ≤2.0 mg/dL (34.2umol/L), AST and ALT≤ 2.5 times the upper limit of normal value, AST and ALT≤ 5 times the upper limit of normal value in patients with liver metastasis.

   B) Kidney: creatinine ≤2.5 mg/dL (221umol/L), creatinine clearance ≥60 mL/min;
9. Understand and sign informed consent to participate in clinical study voluntarily.

Exclusion Criteria:

1. Patients with primary brain tumors other than glioma;
2. Patients with systemic metastasis, poor general condition, and expected survival time less than 1 month;
3. People allergic to pemetrexed;
4. Severe coagulation disorder;
5. Severe active infection and other serious complications;
6. Patients with active viral hepatitis;
7. There are urgent intracranial symptoms (cerebral hernia, etc.), systemic diseases affecting treatment, and basic diseases affecting patients' cognitive function (such as cerebrovascular diseases, Alzheimer's disease, etc.);
8. Pregnant or lactating women;
9. Within 4 weeks prior to enrollment, translumbar administration was performed;
10. Other factors considered by researchers are not suitable candidates.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 24 months
  The percentage of patients with CR and PR in the total number of patients in the same period

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  Frome the starting date of the enrollment until the date of the first documented disease progression or the date of the death from any cause,whichever comes first
Safty(adverse events) | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ren, MD,PhD, Study Chair — Fudan University Pudong Medical Center
Locations (1):
- Fudan University Pudong Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No